CLINICAL TRIAL: NCT04209439
Title: Erector Spinae Plane Block Versus Intravenous Dexketoprofen-trometamol for Treatment of Reno-ureteral Colic: a Randomized Prospective Study
Brief Title: Analgesic Effect of Erector Spinae Plane Block for Renal Colic Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AUTF ANESTHESIAEMERGENCY
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Renal Colic
MeSH Terms: conditions — Renal Colic | interventions — dexketoprofen trometamol

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound guided erector spinae plane block (Active Comparator): 30 ml %0.25 ultrasound-guided erector spinae plane block at the level of T8
  Interventions: Drug: 30 ml %0.25 bupivacaine
- Dexketoprofen-trometamol (Active Comparator): intravenous 50 mg dexketoprofen-trometamol
  Interventions: Drug: Dexketoprofen-trometamol

INTERVENTIONS:
Drug: 30 ml %0.25 bupivacaine — Ultrasound-guided erector spinae plane block
  Arms: ultrasound guided erector spinae plane block
Drug: Dexketoprofen-trometamol — 50 mg Dexketoprofen-trometamol intravenous
  Arms: Dexketoprofen-trometamol

SUMMARY:
Plane blocks have become very popular in recent years with the introduction of ultrasonography into the regional anesthesia and algology practice. Erector spinae plane (ESP) block involves the injection of local anesthetics between erector spinae muscles and transverse process of vertebrae and can block the dorsal and ventral rami of thoracolumbar spinal nerves.

The aim of this study was to evaluate the analgesic efficacy of the erector spine plane block for reno-ureteral colic.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist's physiologic state I-II patients

Exclusion Criteria:

* chronic pain
* bleeding disorders
* renal or hepatic insufficiency
* patients on chronic non-steroidal anti-inflammatory medications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-28 (Actual)

PRIMARY OUTCOMES:
Number of analgesic consumption | 1 hour
  Fentanyl

SECONDARY OUTCOMES:
Numeric Rating Scale | 1 hour
  A NRS involves asking the patient to rate his or her pain from 0 to 10 (11 point scale) with the understanding that 0 is equal to no pain and 10 is equal to worst possible pain. NRS score will be recorded after intervention at 5.,10.,15.,30.,45. and 60. minute

CONTACTS AND LOCATIONS:
Locations (1):
- Ali Ahiskalioglu, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aydin ME, Ahiskalioglu A, Tekin E, Ozkaya F, Ahiskalioglu EO, Bayramoglu A. Relief of refractory renal colic in emergency department: A novel indication for ultrasound guided erector spinae plane block. Am J Emerg Med. 2019 Apr;37(4):794.e1-794.e3. doi: 10.1016/j.ajem.2018.12.042. Epub 2018 Dec 23. PMID 30595427
- [Background] Yayik AM, Ahiskalioglu A, Alici HA, Celik EC, Cesur S, Ahiskalioglu EO, Demirdogen SO, Karaca O, Adanur S. Less painful ESWL with ultrasound-guided quadratus lumborum block: a prospective randomized controlled study. Scand J Urol. 2019 Dec;53(6):411-416. doi: 10.1080/21681805.2019.1658636. Epub 2019 Sep 9. PMID 31496381
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016